CLINICAL TRIAL: NCT03383120
Title: A Randomized Controlled Clinical Trial Comparing Surgical Treatment of Peri-implantitis and Non-surgical Debridement With Adjunctive Diode Laser Therapy
Brief Title: Diode Laser for Treatment of Peri-implantitis
Acronym: LAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Dena Hashim, Principal investigator, University of Geneva, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-02205
Record Dates: First submitted 2017-11-14; First posted 2017-12-26 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Peri-Implantitis; Implant Complication
Keywords: Peri-implantitis; Diode laser; Surgical debridement
MeSH Terms: conditions — Peri-Implantitis | interventions — Laser Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Prospective, single-centre, superiority, randomized, controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: The treatment group will be concealed at all time points from both clinical examiners (N.C., A.Z.) and the biostatistician (D.C.). Only the operator (D.H.) will be aware of the type of treatment to be performed based on the computer-generated allocation table. The un-blinded operator will perform the first follow-up visit one week post-operatively to ensure blinding of the examiners.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser (Experimental): Mechanical debridement of the implant surface using an ultra-sonic device with saline irrigation and plastic curettes, followed by soft tissue curettage using a metallic curette. Adjunctive sub-mucosal diode laser application according to the instructions of the manufacturer (settings: 810 nm, 2.5 W, 50 Hz, 10 ms), 3x for 30 seconds, using a 400-µm thick fiber (Doctor Smile Wiser diode laser, Orcos Medical AG, Küsnacht, Switzerland), will be performed three times at one week intervals (days 0, 7, and 14).
  Interventions: Device: Laser treatment
- Surgery (Active Comparator): Active control includes mechanical debridement of the implant surface using an ultra-sonic device with saline irrigation and plastic curettes, followed by soft tissue curettage using a metallic curette at day 1. An open flap debridement procedure is performed at day 14 using normal saline for implant decontamination. Adjunctive systemic antimicrobials will be prescribed; Amoxi-mepha 500mg 3x/day and Metronidazole 500mg 3x/day, for 1 week. A chlorhexidine 0.2% mouth rinse will also be prescribed 2x/day for one week. Suture removal and prophylaxis are performed 7-10 days post-operatively.
  Interventions: Procedure: Surgical treatment with adjunctive systemic antibiotics

INTERVENTIONS:
Device: Laser treatment — Laser treatment of the peri-implantitis lesion includes mechanical debridement of the implant using an ultrasonic device and plastic curettes followed by diode laser sub-mucosal application for 90 seconds. This is repeated two more times at one-week intervals.
  Other Names: Test
  Arms: Laser
Procedure: Surgical treatment with adjunctive systemic antibiotics — Mechanical debridement of the implant will be done in a similar manner to the test group (without laser application) followed by open flap debridement 2 weeks after, and post-operative prescription of Amoxicillin and Metronidazole systemic antibiotics 3 times per day for a period of 1 week
  Other Names: Control
  Arms: Surgery

SUMMARY:
The primary objective is to evaluate the clinical and patient-centered outcomes of non-surgical mechanical debridement with adjunctive repeated diode laser application (test) in comparison with conventional surgical treatment and adjunctive systemic antibiotics (control), for treatment of peri-implantitis lesions, following an observation period of one year.

DETAILED DESCRIPTION:
Peri-implantitis is a major complication for dental implant patients, with its prevalence estimated in the order of 10% of implants and 20% of patients after 5 to 10 years of implant placement. When left untreated, peri-implantitis may cause progressive tissue destruction, esthetic complications and, eventually, implant loss. Despite numerous clinical trials and systematic reviews, studies have failed to identify a standardized protocol for the treatment of such conditions. Still, current literature and expert opinions recommend mechanical debridement of the implant followed by early evaluation and surgical intervention, implant decontamination using a wide variety of mechanical and chemical methods, then adjunctive systematic antibiotics. However, given the aggressive nature of surgical interventions, the inherent difficulty of decontaminating the implants' rough surfaces with conventional methods, in addition to the growing concerns over antibiotic resistance, the search for alternative approaches has become imperative. Since implant decontamination is the key aspect to resolution of peri-implantitis, different mechanical and chemical methods have been tested in that respect. In recent years, lasers have been attracting significant attention in this particular field. Diode lasers, in particular, have been shown to have potent bactericidal and photobiomodulatory effects promoting wound healing and tissue regeneration. Therefore, the aim of this randomized controlled clinical trial is to evaluate the clinical and patient-centered outcomes of non-surgical debridement with adjunctive repeated diode laser application in comparison with conventional surgical treatment with adjunctive systemic antibiotics for treatment of peri-implantitis lesions following an observation period of one year.

The primary objective is to evaluate the clinical and patient-centered outcomes of non-surgical mechanical debridement with adjunctive repeated diode laser application (test) in comparison with conventional surgical treatment and adjunctive systemic antibiotics (control), for treatment of peri-implantitis lesions, following an observation period of one year.

40 subjects will be randomly distributed into two parallel groups:

1. Test group (n= 20); receiving non-surgical mechanical debridement and adjunctive diode laser application at days 0, 7 and 14.
2. Control group (n= 20); receiving initial mechanical debridement at day 0, followed by open flap debridement and prescription of post-operative systemic antimicrobials at day 14.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* At least one solid screw-type titanium implant diagnosed with peri-implantitis; which is defined as at least one site with probing depth ≥5mm, bleeding on probing and/or suppuration, and radiographic evidence of crater-form bone loss ≥2 threads after insertion of the final prosthetic supra-structure.
* Sound prosthetic supra-structure.

Exclusion Criteria:

* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to Amoxicillin and/or Metronidazole,
* Systemic diseases that could compromise wound healing (i.e. uncontrolled diabetes mellitus, cancer, HIV or bone metabolic disorders), radiation or immunosuppressive therapy,
* Women who are pregnant or breast feeding,
* Known or suspected non-compliance, drug or alcohol abuse,
* Heavy smokers consuming >10 cigarettes/day,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participants not willing to attend regular dental maintenance visits and follow-up evaluations,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Active periodontal disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Resolution of the peri-implantitis | 12 months
  Defined as A absence of probing depths > 4 mm, bleeding on probing or suppuration at the end of the observation period
Types and frequencies of adverse events | 12 months
  Any adverse events related or unrelated to the treatment administered is recorded at the time and appropriate treatment is performed. The frequency, duration and intensity is also recorded.
Patient reported outcomes at 1 week | 1 week post-operatively
  A visual analogue scale is used to evaluate post-operative discomfort and patient's perception of the administered treatment 1 week post-operatively.The scale measures a total of 100 mm ranging between 0-100; 0 indicating absence of pain and 100 being the worst pain imaginable.
Patient reported outcomes at 12 months | 12 months
  A visual analogue scale is used to evaluate general patient's perception of the administered treatment 12 months post-operatively.The scale measures a total of 100 mm ranging between 0-100; 0 indicating lack of discomfort or pain and complete satisfaction and 100 being completely unsatisfied and/or with persisting pain or other symptoms.

SECONDARY OUTCOMES:
Change in marginal bone levels | 12 months
  Changes in peri-implant marginal bone levels are measured on intra-oral radiographs taken at baseline and 12 months post-operatively. Two independent examiners perform measurements and mean values are taken. This outcome is only calculated 12 months postoperatively.
Differences between groups regarding changes in mean marginal bone level changes | 12 months
  Comparison in mean marginal bone level changes (outcome 4) are performed between the test and control groups
Number of residual pockets > 4 mm | 12 months
  Number of residual peri-implant pockets exceeding 4 mm are measured around all included implants at the end of the observation period to asses the presence of any residual peri-implant soft-tissue inflammation
Changes in probing depth | 12 months
  The change in mean probing depth between baseline and 12 months is calculated to assess treatment outcomes and disease resolution around all included implants. This outcome is calculated only once 12 months post-operatively.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Geneva, Geneva, Genève 4, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided